CLINICAL TRIAL: NCT06765564
Title: Clinical Study of Human Induced Pluripotent Stem Cells Derived Motor Neuron Precursor(iPSC-MNP) Cells for the Treatment of Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Clinical Study of Induced Pluripotent Stem Cells Derived Motor Neuron Precursor Cell Therapy for Amyotrophic Lateral Sclerosis (ALS)
Acronym: iPSC-MNP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XS2022002
Record Dates: First submitted 2023-11-13; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: ALS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One-arm study (Experimental): Use of experimental drug
  Interventions: Drug: iPSC-MNP

INTERVENTIONS:
Drug: iPSC-MNP — Using iPSC-MNP Cells for the Treatment of ALS Patients

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a severe neurodegenerative disease in the human motor system characterized by the selective involvement of spinal cord anterior horn cells, brainstem motor nuclei, and the corticospinal tract. It predominantly presents as concurrent damage to upper and lower motor neurons.

Induced pluripotent stem cells (iPSCs) are a type of induced pluripotent stem cell derived from autologous or allogeneic cell sources. They can differentiate into various functional cell types, including specific motor neuron cells. iPSCs are used for stem cell replacement therapy. iPSCs hold significant clinical potential for ALS treatment. The iPSC database with human leukocyte antigen characteristics may represent a promising technology. This technology has the potential to obtain high-quality cell products and reduce the risk of graft rejection. Moreover, human iPSCs have demonstrated a certain degree of efficacy in the transplantation of neural stem/progenitor cells derived from ALS rodent models.

The potential mechanisms of iPSC therapy for ALS include: the differentiated motor neuron precursor cells can replace damaged motor neurons, and restore motor conduction function; by secreting neurotrophic factors, they protect neurons; through immune regulation, they inhibit inflammatory reactions, and slow the progression of ALS.

Xellsmart Biomedical (Suzhou) Co., Ltd. is developing an injectable solution for ALS treatment using human iPSC-derived motor neuron precursor cells to address the pressing need for ALS therapy.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, multiple-dose, investigator-initiated interventional clinical trial aimed at preliminary exploring the safety of the investigational drug. The study is divided into three phases: a baseline period (7 days), a treatment period (45 days), and a follow-up period (6 months).

Baseline Period: The ALS subjects need to sign the informed consent form for the clinical trial (including the installation surgery for the Sofia drug pouch) and undergo baseline assessments before the transplant surgery to exclude any conditions that would disqualify them from participation. The subjects need to undergo medical history collection, vital signs and physical examinations, laboratory tests, various other auxiliary examinations, and perform self-assessment of their physical condition. The investigator records clinical symptoms, scores and records various scales and tables. [including ALS Functional Rating Scale-Revised (ALSFRS-R), Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Hamilton Depression Rating Scale (HAMD 17), Hamilton Anxiety Rating Scale (HAMA), Fatigue Severity Scale (FSS)]. Qualified subjects will subsequently take oral immunosuppressants for three months, and the clinical research investigator will adjust the dosage and medication duration based on the subjects' rejection response and tolerability.

Treatment Period: At Day -3 of the treatment period, the surgical expert administers general anesthesia to the subjects and, under the guidance of a robot, installs the Sofia drug pouch. On the first day post-surgery, through head CT and other examinations, adverse events (AEs and SAEs) are assessed. On Treatment Day 0 (i.e., 3 days post-surgery), the first stem cell transplantation begins. Subjects undergo vital sign monitoring, physical examinations, and record self-assessments of their physical condition and clinical symptoms before undergoing intraventricular stem cell transplantation. The investigator injects 2 mL of human iPSC-derived motor neuron precursor cells (5×107 cells) through the subcutaneous drug pouch. Subsequently, the same dose of stem cells is administered through the drug pouch every half month, totaling four times. After the administration, subjects are advised to lie flat for one hour, with simultaneous monitoring of vital signs and blood oxygen saturation, and recording of any possible adverse events (AEs and SAEs). On the third day after each stem cell transplantation treatment, subjects undergo safety assessments (vital signs, physical examinations, laboratory tests, 12-lead electrocardiogram, cerebrospinal fluid routine, ultrasound, and imaging examinations, etc.) and an evaluation of the impact of this study on the efficacy of individual ALS subjects (patient self-assessment of condition and clinical symptoms, scales [ALSFRS-R, MMSE, MoCA, HAMD 17, HAMA, FSS], electrophysiological parameter testing, FVC, and cerebrospinal fluid neurotrophic factor detection).

Follow-up Phase: Subjects return to the clinical research center for safety and effectiveness assessments at 1 month, 3 months, and 6 months after finishing all the stem cell transplantations (i.e., 2.5 months, 4.5 months, and 7.5 months after the first stem cell transplantation). For subjects who do not complete all four stem cell transplantations, the follow-up schedule is adjusted based on the completion time of the stem cell transplantation. For safety reasons, the next subject can only be enrolled after the previous subject has completed the stem cell transplantation and been observed for 6 months without the occurrence of acute or delayed SAEs. The clinical research center should be equipped to handle unexpected acute, severe adverse events, such as allergic reactions and medication-related reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients themselves or their legal guardians must consent to undergo this treatment protocol and sign the Informed Consent Form (ICF).
2. Age between 18 and 60 years, inclusive, with no gender restrictions.
3. Diagnosed with ALS according to the World Federation of Neurology criteria, and the initial diagnosis date is between 6 to 24 months before the screening date.
4. Patients who have received standard treatment in the past with poor efficacy or disease progression.
5. Forced Vital Capacity (FVC) should be ≥50%.
6. During any night of the screening period, the total time with peripheral blood oxygen saturation <90% should not exceed 2%.
7. Patients should be deemed by the investigator to be in good nutritional status, with a Body Mass Index (BMI) ≥18.5.
8. Male patients and their spouses, as well as women of childbearing age, should agree to implement effective contraceptive measures from the time of signing the ICF until one year after the start of treatment.
9. Patients should be able to cooperate in the collection and preservation of medical history data and the visit process.

Exclusion Criteria:

1. Patients with symptoms of neuromuscular weakness but cannot be conclusively determined to have ALS.
2. Patients diagnosed with severe cognitive impairment, clinical dementia, or major psychiatric disorders, including but not limited to schizophrenia, bipolar disorder, or severe depression, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
3. Patients with any disease that impairs nerve or muscle function, such as peripheral neuropathy or metabolic myopathy.
4. Patients with a history of malignant tumors or a previous diagnosis of malignancy.
5. Within the two weeks preceding the screening period, patients who experienced acute active infections requiring treatment with antibiotics, antiviral drugs, or antifungal medications.
6. ALS patients with concomitant respiratory failure.
7. Patients who have previously undergone any allogeneic cell therapy or organ transplantation.
8. Patients who have Participated in other clinical trials within the three months prior to screening.
9. Patients with a history of tracheostomy or those using mechanical ventilatory support.
10. Patients with a documented history of severe allergic reactions to general anesthesia drugs or previous severe allergic reactions for other reasons.
11. Patients with intracranial organic diseases causing increased intracranial pressure.
12. Patients with elevated liver function test results during the screening period, such as total bilirubin >1.5 times the upper limit of normal (ULN), or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times ULN.
13. Patients who have abnormal kidney function test results during the screening period, such as serum creatinine >1.5 mg/dL or an estimated creatinine clearance rate <60 mL/min calculated by the Cockcroft and Gault formula.
14. Other clinically significant laboratory abnormalities during the screening period.
15. Patients with hepatitis A, active hepatitis B (HBsAg positive and HBV DNA ≥500 IU/ml, excluding drug- or other-caused hepatitis), active hepatitis C (anti-HCV antibody positive and HCV RNA positive), hepatitis E, human immunodeficiency virus (HIV) antibody positive, or syphilis treponemal antibody positive.
16. Patients with impaired consciousness.
17. Coagulation abnormalities (prothrombin time [PT] or international normalized ratio [INR] >1.5 times ULN; activated partial thromboplastin time [APTT] >1.5 times ULN) or those currently receiving anticoagulation therapy.
18. Poorly controlled hypertension, with systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg after treatment.
19. Severe diabetes with late complications; patients with other diseases affecting limb mobility (e.g., limping, osteoarthritis, rheumatoid arthritis, gout, etc.).
20. Patients who have undergone surgery or experienced trauma (including fractures) in the past month.
21. Pregnant or breastfeeding women.
22. Patients who, in the opinion of the investigator, have poorly controlled systemic diseases or other conditions that make them unsuitable for participation in this clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-03-13 (Estimated); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse event (AE) and serious adverse event(SAE) | 0、1、3、6 month
  AE occurring throughout the study period will be evaluated using the CTCAE V5.0 standard.
  AE/SAE were evaluated by laboratory examination and imageological examination, measuring method：
  1. Head MRI, whole spine MRI, chest CT examination;
  2. Changes in vital signs, 12-lead electrocardiogram, ultrasound (thyroid, abdomen, heart, genitourinary system) examination, and neurological signs;
  3. Changes in blood routine, urine routine, stool routine, finger end blood oxygen saturation, serum immunoglobulin, cerebrospinal fluid routine, liver function, kidney function, electrolyte, muscle enzyme, lipid, blood glucose, glycated hemoglobin, coagulation function, tumor markers, various hepatitis viruses, treponema lutei antibodies, HIV antibodies and other indicators.

SECONDARY OUTCOMES:
effective of Induced Pluripotent Stem Cells Derived Motor Neuron Precursor Cell | 0、1、3、6 month
  ALS functional assessment: Changes in ALSFRS-R scale score; The ALSFRS-R includes 12 different tasks designed to provide a representative picture of the physical abilities most commonly affected by ALS. These tasks include speaking, salivation, swallowing, writing, climbing stairs, turning in bed, walking, dressing and hygiene, and three different measures of respiratory capacity. Each task is rated on a scale of 0 to 4-0 indicates the inability to perform the task, and 4 indicates the ability to perform it without difficulty. These ratings are then summed to yield a total score ranging from 0 to 48, with 0 being the worst and 48 being the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Shang hai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided